CLINICAL TRIAL: NCT03413072
Title: Galectin-3 as a Predictor for Thromboembolic Formation in Patients With Non Valvular Atrial Fibrillation Assessed by CHA₂DS₂-VASc Scoring
Brief Title: Galectin-3 for Thromboembolic Formation in Patients With Atrial Fibrillation CHA₂DS₂-VASc Scoring
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Fatma El-sayed Moustafa, principal investigator, Assiut University
Other Study IDs: G-3A
Record Dates: First submitted 2018-01-16; First posted 2018-01-29 (Actual); Last update posted 2018-01-29 (Actual); Status verified 2018-01

CONDITIONS: Atrial Fibrillation; Stroke
MeSH Terms: conditions — Atrial Fibrillation; Stroke

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Atrial Fibrillation is considered as one of a common cardiac arrhythmia that presented with rapid and irregular rhythm and has an increased incidence.There are different types of atrial fibrillation one of these is paroxysmal atrial fibrillation that defined as lasts longer than 30 seconds and lasting less than 7 days, while atrial fibrillation lasting more than 7 days to less than one year or requiring pharmacological or electrical cardioversion is called persistent atrial fibrillation, referring to the American Heart Association 2006 guidelines.Patients with atrial fibrillation suffer from serious complications like stroke due to thromboembolism, heart failure and death. Risk of stroke is 5-folds in patients with atrial fibrillation in addition to presence or absence of another clinical risk factors.

DETAILED DESCRIPTION:
In 2001, the CHADS₂ score (congestive heart failure, hypertension, age ≥75 years, diabetes mellitus, stroke) was developed to predict the risk of stroke in patients with non rheumatic atrial fibrillation.In this score, each patient giving one point for congestive heart failure , hypertension , age equal or more than 75 years, diabetes mellitus and two points for stroke, transient ischemic attack.

In 2010, CHADS₂ was expanded to include three additional independent risk factors: vascular disease (coronary artery disease, peripheral artery disease, aortic atherosclerosis), age 65-74 years, and female sex. So new, more inclusive scoring system is the CHA₂DS₂-VASc. Each patient giving one point for congestive heart failure, hypertension, diabetes mellitus, vascular disease, age 65-74 and female gender and two point for history of stroke, transient ischemic attack and age≥75.

The CHA₂DS₂-VASc score is better to predict stroke risk in non valvular atrial fibrillation patients with a baseline CHADS₂ score of 0 to 1. The 2014 American Heart Association/ American College of Cardiology/ Heart Rhythm Society guidelines also recommend the CHA₂DS₂-VASc for stroke risk in patients with non valvular atrial fibrillation. The 2016 European Society of Cardiology guidelines recommend using the CHA₂DS₂-VASc score to predict stroke risk in atrial fibrillation patients and to give oral anticoagulants to men with a score of 1 or higher and women with a score of 2 or higher.

Stroke is a serious vascular problem, 25-30 percent of the cause is atrial fibrillation inspite of paroxysmal or persistent types.

Galectin-3 is known as a soluble beta-galactoside binding lectin that secreted by immune cell and mediates profibrotic pathways. Also it has a role in inflammation, cell proliferation, and tissue repair. So, it is involved in multiple diseases as liver, kidney, inflammatory disease.

In cardiac disease, it has a role in pathophysiology of atrial fibrillation, heart failure, myocardial infarction as the level is found high in patients with ST segment elevation myocardial infarction than normal persons and according to the level the outcome of disease is suggested.

Also if galectin-3 is greater than the median level, the patients have a higher risk of new or recurrent heart failure. Galectin-3 has been approved by the Food and Drug Administration as a prognostic biomarker in congested heart failure to be used in conjunction with clinical evaluation.

Galectin-3 has an ability of binding to von willbrand factor so help in modulation of early thrombus formation, as the glycans on human factor VIII are similar to von willbrand factor.

ELIGIBILITY:
Inclusion Criteria:

1. Gender: men and women.
2. Age >18 years.
3. Diagnosed as non valvular atrial fibrillation patients either paroxysmal or persistent types.

Exclusion Criteria:

1. pregnancy
2. valvular heart diseases.
3. Congenital heart diseases.
4. Heart failure.
5. Ischemic heart disease.
6. Inflammatory diseases.
7. Cancer.
8. Thyroid disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with non valvular atrial fibrillation either paroxysmal or persistent types above 18 years.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2018-06 (Estimated); Primary Completion 2019-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Correlation of Galectin-3 blood Level with the risk of thromboembolic complications among patients with paroxysmal and persistent atrial fibrillation as assessed by CHA₂DS₂-VASc scoring. | one year

SECONDARY OUTCOMES:
Correlation of the level of galectin-3 in the blood with changes in activated partial thromboplastin time | One year

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wolf PA, Abbott RD, Kannel WB. Atrial fibrillation as an independent risk factor for stroke: the Framingham Study. Stroke. 1991 Aug;22(8):983-8. doi: 10.1161/01.str.22.8.983. PMID 1866765
- [Background] Magnani JW, Rienstra M, Lin H, Sinner MF, Lubitz SA, McManus DD, Dupuis J, Ellinor PT, Benjamin EJ. Atrial fibrillation: current knowledge and future directions in epidemiology and genomics. Circulation. 2011 Nov 1;124(18):1982-93. doi: 10.1161/CIRCULATIONAHA.111.039677. PMID 22042927
- [Background] Lip GY, Nieuwlaat R, Pisters R, Lane DA, Crijns HJ. Refining clinical risk stratification for predicting stroke and thromboembolism in atrial fibrillation using a novel risk factor-based approach: the euro heart survey on atrial fibrillation. Chest. 2010 Feb;137(2):263-72. doi: 10.1378/chest.09-1584. Epub 2009 Sep 17. PMID 19762550
- [Background] Chao TF, Liu CJ, Chen SJ, Wang KL, Lin YJ, Chang SL, Lo LW, Hu YF, Tuan TC, Wu TJ, Chen TJ, Tsao HM, Chen SA. Atrial fibrillation and the risk of ischemic stroke: does it still matter in patients with a CHA2DS2-VASc score of 0 or 1? Stroke. 2012 Oct;43(10):2551-5. doi: 10.1161/STROKEAHA.112.667865. Epub 2012 Aug 7. PMID 22871677
- [Background] Henderson NC, Mackinnon AC, Farnworth SL, Poirier F, Russo FP, Iredale JP, Haslett C, Simpson KJ, Sethi T. Galectin-3 regulates myofibroblast activation and hepatic fibrosis. Proc Natl Acad Sci U S A. 2006 Mar 28;103(13):5060-5. doi: 10.1073/pnas.0511167103. Epub 2006 Mar 20. PMID 16549783
- [Background] McCullough PA, Olobatoke A, Vanhecke TE. Galectin-3: a novel blood test for the evaluation and management of patients with heart failure. Rev Cardiovasc Med. 2011;12(4):200-10. doi: 10.3909/ricm0624. PMID 22249510
- [Background] O'Sullivan JM, Jenkins PV, Rawley O, Gegenbauer K, Chion A, Lavin M, Byrne B, O'Kennedy R, Preston RJ, Brophy TM, O'Donnell JS. Galectin-1 and Galectin-3 Constitute Novel-Binding Partners for Factor VIII. Arterioscler Thromb Vasc Biol. 2016 May;36(5):855-63. doi: 10.1161/ATVBAHA.115.306915. Epub 2016 Mar 24. PMID 27013611